CLINICAL TRIAL: NCT00906282
Title: Phase II Trial of Preoperative Pemetrexed and Carboplatin in Patients With Select Stage IB, II, and III Non-Squamous Non-Small-Cell Lung Cancer
Brief Title: Preoperative Pemetrexed and Carboplatin for Select Stage IB, II, and III Non-Squamous Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 186
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: neoadjuvant NSCLC; NSCLC; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pemetrexed/Carboplatin (Experimental): 4 cycles of preoperative treatment (1 Cycle = 21 days):
  Pemetrexed: 500 mg/m2 intravenously (IV) for 10 minutes on Day 1 each cycle; Carboplatin: AUC 6.0 by IV on Day 1 each cycle.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 IV over 10 minutes on Day 1 of every 3-week treatment cycle for a total of 4 cycles (12 weeks).
  Other Names: Alimta
Drug: Carboplatin — AUC 6.0 IV on Day 1 of every 3-week treatment cycle for a total of 4 cycles (12 weeks).
  Other Names: 41575-94-4

SUMMARY:
The purpose of this multi-center Phase II trial is to examine the impact of pemetrexed/carboplatin in the preoperative treatment of patients with select stage IB, II,and III non-squamous NSCLC. Because patients with non-squamous type NSCLC have been shown to have better survival rates than patients with squamous tumors when given pemetrexed with a platinum agent, only patients with non-squamous NSCLC (adenocarcinoma, large cell, and undifferentiated), not including squamous histology, will be allowed to participate in this study. If this novel regimen proves to be safe and active in this setting, it will provide rationale for further investigation in a larger, prospective, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed NSCLC (adenocarcinoma, large cell, and undifferentiated). Patients with squamous histology are not eligible.
2. Life expectancy of at least 12 weeks.
3. Patients with the following stages of NSCLC:

   * T2 N0 tumors: Limited to tumors >=4 cm.
   * T1-2 N1 tumors.
   * T3 N0-1 tumors (excluding superior sulcus tumors): Including tumors involving the chest wall, proximal airway, or mediastinal pleura where preoperative radiotherapy is not planned.
   * T1-2 N2 tumors: For patients with N2 disease involving one zone (Upper zone (R), AP zone (L), subcarinal zone, or lower zone) and nodes <=2cm in diameter.
   * T4 N0-1 tumors (excluding superior sulcus tumors): T4 lesions other than malignant effusions where radiotherapy is not planned.
4. Patients with clinical N2 involvement must have histologic confirmation by mediastinoscopy (or alternate biopsy procedure).
5. Tumors should be considered potentially resectable.
6. No evidence of extrathoracic metastatic disease.
7. Patients must have measurable disease by RECIST criteria.
8. Patients must be candidates (medically) for chemotherapy followed by surgical resection.
9. Adequate recovery from recent surgery. At least 1 week must have elapsed from the time of a minor surgery; at least 3 weeks must have elapsed from the time of a major surgery.
10. Laboratory values as follows:

    * Absolute neutrophil count (ANC) >=1500/μL
    * Hemoglobin (Hgb) >=10 g/dL
    * Platelets >=100,000/uL
    * AST/SGOT and ALT/SGPT within normal limits (WNL)
    * Total bilirubin within normal limits (WNL)
    * Calculated creatinine clearance >=45 mL/min
11. ECOG Performance Status grade 0 or 1.
12. The ability to interrupt NSAIDS 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of Alimta.
13. The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.
14. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
15. Patient must be accessible for treatment and follow-up.
16. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Patients with the following stages are excluded:

   * T1 N0;
   * T2 N0, with primary tumor <4 cm;
   * T1-2 N2, with multiple zones of N2 involvement;
   * T3-4 N2;
   * Any N3;
   * Any TxNxM1 disease; or
   * Any stage where surgery and/or chemoradiotherapy is the preferred initial approach in management, as deemed by the treating physician.
2. Squamous or predominant squamous mixed histologies.
3. Mixed small-cell and non-small cell histologies.
4. Pulmonary carcinoid tumors.
5. Presence of third space fluid which cannot be controlled by drainage.
6. Use of erythropoietin as a hematopoietic growth factor is not allowed.
7. Cardiac disease, including: congestive heart failure (CHF) > Class II per New York Heart Association (NYHA) classification; unstable angina (anginal symptoms at rest) or new-onset angina (i.e., began within the last 3 months), or myocardial infarction within the past 6 months; symptomatic CHF, unstable angina pectoris, cardiac arrhythmia, or cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
8. Women who are pregnant (positive pregnancy test) or lactating.
9. Use of any non-approved or investigational agent within 30 days of administration of the first dose of study drug.
10. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
11. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
13. History of hypersensitivity to active or inactive excipients of any component of treatment.
14. Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (12):
- United States (12):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Oncology Hematology Care, Cincinnati, Ohio
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Aug 2009 and Jul 2013, 46 patients with potentially resectable non-squamous NSCLC were enrolled from 10 participating sites in the U.S.
Pre-assignment Details: Patients (pts) received up to 4 cycles (12 weeks) of preoperative chemotherapy and were restaged after 6 and 12 weeks. Pts with progressive disease or intolerable toxicity came off study; pts who remained surgical candidates had resection at weeks 15-18. Following resection pts received no further planned protocol treatment.
Groups:
- Pemetrexed/Carboplatin/Surgery: Up to 12 weeks of preoperative chemotherapy:
  * Pemetrexed: 500 mg/m2 intravenously (IV) for 10 minutes on Day 1 each cycle;
  * Carboplatin: AUC 6.0 by IV over 30-60 minutes on Day 1 each cycle
  Weeks 15-18: Patients deemed surgical candidates will have resection.
Period: Preoperative Chemotherapy
Arm/Group | Pemetrexed/Carboplatin/Surgery
Started | 46
Completed | 27 (2 of 27 patients completed less than 4 cycles and were deemed surgical candidates.)
Not Completed | 19
Not completed — Withdrawal by Subject | 2
Not completed — Not surgical candidates, off study | 10
Not completed — Progressive disease | 6
Not completed — Toxicity | 1
Period: Surgical Resection
Arm/Group | Pemetrexed/Carboplatin/Surgery
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed/Carboplatin/Surgery: Up to 12 weeks (4 cycles) of preoperative treatment given on Day 1 of each 21-day cycle:
  * Pemetrexed: 500 mg/m2 intravenously (IV) over 10 minutes
  * Carboplatin: AUC 6.0, IV infused over 30-60 minutes
  At weeks 15-18, surgical candidates will have resection.
Arm/Group | Pemetrexed/Carboplatin/Surgery
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 65 [42 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 28
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 42
  African-American | 4
Region of Enrollment [Number; unit: participants]
  United States | 46
Clinical Stage of Cancer [Number; unit: participants] — Number of patients based on clinical stage of disease at study entry.
  participants
    Stage 1B | 5
    Stage IIA/II/B | 17
    Stage IIIA | 23
    Stage IIIB | 1

OUTCOME MEASURES:

1. Primary Outcome: 3-Year Overall Survival Rate
Description: The percentage of patients who were alive at 3 years from time of first study treatment until date of death from any cause. Overall survival is shown for the Intent-to-Treat population.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed/Carboplatin/Surgery
Number analyzed (Participants) | 46
percentage of participants | 45 [30 to 60]

2. Secondary Outcome: Objective Tumor Response
Description: Objective Tumor Response defined as the percent of patients who completed up to 4 cycles of pre-operative chemotherapy and achieved a complete response (CR) or partial response (PR) assessed by Response Evaluation in Solid Tumors (RECIST) 1.0. Patients with stable disease (SD) or response to treatment were deemed surgical candidates. [CR=disappearance of all target tumors; PR= ≥30% decrease in the sum of the longest diameters of target tumors. SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.]
Time Frame: At 6 and 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed/Carboplatin/Surgery
Number analyzed (Participants) | 46
percentage of participants
  PR | 41
  SD | 48

3. Secondary Outcome: Pathologic Response Rate
Description: Percent of patients having a pathological complete or partial response (pCR or pPR) at surgery. pCR defined as complete removal of all tumor. pPR defined as residual viable tumor demonstrated in the resected specimen.
Time Frame: weeks 15 -18
Measure: Number; unit: percentage of participants
Arm/Group | Pemetrexed/Carboplatin/Surgery
Number analyzed (Participants) | 27
percentage of participants
  pPR | 100
  pCR | 0

4. Secondary Outcome: Rate of Residual Disease as an Assessment of Pathological Partial Response (pPR)
Description: pPR was further assessed by the amount of residual tumor measured at surgery: microscopic residual disease = less than 1 centimeter (<1 cm); macroscopic residual disease = 1 centimeter or greater (≥1 cm).
Time Frame: At 15-18 weeks
Population: The amount of residual tumor measured in centimeters (cm).
Measure: Median (Full Range); unit: centimeters
Arm/Group | Pemetrexed/Carboplatin/Surgery
Number analyzed (Participants) | 27
centimeters | 2.5 [0.5 to 9.5]

5. Secondary Outcome: Complete Resection Rate
Description: The percent of patients who had surgical resection listed by procedure type: lobectomy or pneumonectomy, or resection of adjacent chest wall or mediastinal structures when appropriate. Surgery followed standard guidelines for resection of non-small-cell lung cancer (NSCLC).
Time Frame: At weeks 15-18
Measure: Number; unit: percentage of patients
Groups:
- Pemetrexed/Carboplatin/Surgery: Up to 12 weeks (4 cycles) of preoperative treatment on Day 1 of each 21-day cycle:
  * Pemetrexed: 500 mg/m2 intravenously (IV) over 10 minutes
  * Carboplatin: AUC 6.0, IV infused over 30-60 minutes
  At weeks 15-18, surgical candidates will have resection.
Arm/Group | Pemetrexed/Carboplatin/Surgery
Number analyzed (Participants) | 27
percentage of patients
  Lobectomy | 70
  Wedge Resection | 15
  Pneumonectomy | 11
  Bilobectomy | 4

ADVERSE EVENTS:
Time Frame: Every 3 weeks up to 12 weeks during preoperative treatment, then every 3 months post surgery for years 1-2, and every 6 months thru years 3-5..
Groups:
- Pemetrexed/Carboplatin: All patients who received at least 1 dose of study treatment were included in the safety analysis.
Arm/Group | Pemetrexed/Carboplatin
Serious Adverse Events (participants affected / at risk) | 18/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed/Carboplatin (N=46)
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Anorectal cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count (Investigations) | 1
Platelet count decreased (Investigations) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed/Carboplatin (N=46)
Anaemia (Blood and lymphatic system disorders) | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 22
Leukopenia (Blood and lymphatic system disorders) | 17
Neutropenia (Blood and lymphatic system disorders) | 18
Lymphopenia (Blood and lymphatic system disorders) | 4
Fatigue (General disorders) | 36
Oedema Peripheral (General disorders) | 5
Pyrexia (General disorders) | 6
Mucosal Inflammation (General disorders) | 5
Asthenia (General disorders) | 3
Chest pain (General disorders) | 3
Chills (General disorders) | 3
Nausea (Gastrointestinal disorders) | 29
Constipation (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Haemoglobin (Investigations) | 9
Platelet count decreased (Investigations) | 4
Platelet count (Investigations) | 8
Neutrophil count (Investigations) | 8
Neutrophil count decreased (Investigations) | 5
Weight decreased (Investigations) | 6
White blood cell count (Investigations) | 5
Haemoglobin decreased (Investigations) | 4
Blood creatinine decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Blood glucose increased (Investigations) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 8
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Insomnia (Psychiatric disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.